CLINICAL TRIAL: NCT06957171
Title: Correlation Between Intraoperative Fluid Volume and Postoperative Inferior Vena Cava Distensibility Index in Pediatric Operations
Brief Title: Assess the Potential of the IVC Distensibility Index as a Predictor of Postoperative Fluid Status in Children.
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MS 728/2024
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Intraoperative Fluid Volume; Inferior Vena Cava Diameter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1: Age 1-4 years, Conservative Fluid: Patients aged 1 to 4 years receiving intraoperative fluid <10 ml/kg/h.
- Group 2: Age 1-4 years, Liberal Fluid: Patients aged 1 to 4 years receiving intraoperative fluid ≥10 ml/kg/h.
- Group 3: Age 4-8 years, Conservative Fluid: Patients aged 4 to 8 years receiving intraoperative fluid <10 ml/kg/h.
- Group 4: Age 4-8 years, Liberal Fluid: Patients aged 4 to 8 years receiving intraoperative fluid ≥10 ml/kg/h.
- Group 5: Age 8-12 years, Conservative Fluid: Patients aged 8 to 12 years receiving intraoperative fluid <10 ml/kg/h.
- Group 6: Age 8-12 years, Liberal Fluid: Patients aged 8 to 12 years receiving intraoperative fluid ≥10 ml/kg/h.

SUMMARY:
The investigators will assess the relationship between the amount of fluid administered during pediatric surgery and the subsequent IVC distensibility index postoperatively.

DETAILED DESCRIPTION:
Preoperative settings:

Preoperative assessment will be done which includes Medical History and Clinical Examination: Age, gender, and weight will be recorded, Number of fasting hours, Surgical History documentation of previous surgeries, if any, including details on anesthetic techniques. family history of cardiovascular, renal, or fluid balance disorders. Information on any known allergies, particularly to medications, as well as a list of current medications being taken by the patient. Any coexisting medical conditions, particularly autoimmune, inflammatory, or chronic diseases, will be documented (e.g., asthma, diabetes, renal insufficiency).

Specific Examination for IVC Distensibility:

• Ultrasonographic Examination: Preoperative ultrasound will be used to measure the baseline Inferior Vena Cava (IVC) diameter and assess its distensibility as a part of the preoperative evaluation.

Preoperative Assessment of Fluid Balance:

• Laboratory Tests: Baseline blood tests, including complete blood count, serum electrolytes, and renal function tests, will be performed to assess overall fluid and electrolyte balance.

Intraoperative Monitoring:

Intraoperative fluid strategy will be followed with the local protocol 10 ml/kg/h will be given, and additional boluses 10-20 ml/kg if needed (in case of hemodynamic instability, increasing lactate), losses will be compensated with fluid or blood (if exceeded the allowable blood loss).

This fluid regimen is individualized by the attending anaesthesiologist according to the actual requirement, The volume of fluids administered intraoperatively will be meticulously recorded. Urine Output Documentation of baseline urine output as an indicator of renal function and fluid status.

Postoperative Settings:

All ultrasonographic measurments of IVC will be performed at the end of surgery, before extubation (patient is anaesthetized and completely relaxed, in the supine position, PEEP less than 7 cmH2O and tidal volume 6-8 ml/kg The probe will be placed at the sub xiphoid area and measurements will be obtained in M-mode imaging performed 2 to 3 cm distal to the right atrium in the long-axis subcostal view..IVC diameter during inspiration (IVCi) and expiration (IVCe) will be measured, Collapsibility index (CI) measured as difference between IVCe, IVCi divided on IVCe (CI = IVCe - IVCi /IVCe x100).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 1-12 years.
* ASA status I - II
* Patients undergoing elective surgical procedures requiring general anesthesia.

Exclusion Criteria:

* Patients with known congenital heart disease, valvular heart disease or Pulmonary hypertension

  * Renal disorders (Acute or Chronic).
  * PEEP more than 7 cmH2O at time of assessment of IVC distensibility index

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include pediatric patients aged 1-12 years undergoing elective surgery under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Inferior Vena Cava distensibility index | At the end of surgery, before extubation
  All ultrasonographic measurments of IVC will be performed at the end of surgery, before extubation (patient is anaesthetized and completely relaxed, in the supine position, PEEP less than 7 cmH2O and tidal volume 6-8 ml/kg The probe will be placed at the sub xiphoid area and measurements will be obtained in M-mode imaging performed 2 to 3 cm distal to the right atrium in the long-axis subcostal view..IVC diameter during inspiration (IVCi) and expiration (IVCe) will be measured, Collapsibility index (CI) measured as difference between IVCe, IVCi divided on IVCe (CI = IVCe - IVCi /IVCe x100).

CONTACTS AND LOCATIONS:
Overall Officials: Rawan Abu Deif, M.B.B.CH, Principal Investigator — Anaesthesia resident Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before 1/2026
Access Criteria: Free